CLINICAL TRIAL: NCT03277612
Title: Effects of C-section Delivery on Infant Brain Development
Status: Terminated | Type: Observational
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206515
Record Dates: First submitted 2017-06-28; First posted 2017-09-11 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, stool, vaginal swabs, and breast milk samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C-Section: Infants delivered by C-section
- Vaginal Delivery: Infants delivered by spontaneous vaginal delivery after C-section.

SUMMARY:
The study will help investigators learn more about whether different delivery modes influence infant's brain development

DETAILED DESCRIPTION:
For this study, the investigators are enrolling women who are pregnant with their second child who are planning to have a planned C-section or a spontaneous vaginal birth after C-section. The investigators will see the pregnant mom at 36 weeks pregnant and then have the mom and the baby return for a visit at 2 weeks postnatal.

ELIGIBILITY:
Inclusion Criteria:

* Conceived without fertility treatments
* Singleton pregnancy recruited at or before 36 weeks of gestation
* Second parity with planned repeated C-section delivery or with planned spontaneous vaginal delivery after C-section.

Exclusion Criteria:

* Preexisting medical conditions
* Sexually transmitted diseases
* Medical complications developed during pregnancy
* Medical complications developed during labor and delivery
* Emergency c-section delivery
* Infants born preterm or post-term
* Infants needing mechanical ventilation, have congenital abnormalities, birth defects, intrauterine growth restriction, low Apgar score (<7), or other medical issues developed at birth or before 2 weeks of age affecting the outcome of interest as determined by the PI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and their unborn child
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome and how it effects Brain Structure | up to 2 weeks
  Evaluate the relationship between gut microbiome and brain structural in infants based on mode of delivery as determined by an MRI
Gut Microbiome and how it effects brain function | up to 2 weeks
  Evaluate the relationship between gut microbiome and brain function in infants based on mode of delivery as determined by an MRI

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Ou, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No